CLINICAL TRIAL: NCT07198022
Title: Comparative Evaluation of Application of Topical Anesthetic Gel, Solution and Cryotherapy
Brief Title: Cryotherapy as a Topical Anesthetic in Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Bilal OZMEN, Assoc.Prof.Bilal OZMEN, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024000316
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Topical Anesthesia; Pediatric Dentistry; Cryotherapy
Keywords: topical anesthetic; cryotherapy; injection; children
MeSH Terms: interventions — Cryotherapy; Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Topical Anesthetic Solution (Active Comparator): In spray group, as a topical anaesthetic solution containing 10% lidocaine will be applied to the injection site with the help of a pressel for 20 seconds after the application area is dried by squeezing a cotton pellet. The taste/odour evaluation of the applied topical anaesthetic material will be measured with the 3 Category Hedonic Scale. After sufficient numbness is achieved, local infiltrative injection will be performed. Anxiety levels will be evaluated by measuring with the same parameters before topical anaesthesia application, during topical anaesthesia application and injection.
  Interventions: Drug: topical anesthetic
- Topical Anesthetic Gel (Experimental): In topical anesthetic gel group, a gel containing %20 benzocain with strawberry aroma, will be applied to the injection site with the help of a pressel for 20 seconds after the application area is dried by squeezing a cotton pellet. The taste/odour evaluation of the applied topical anaesthetic material will be measured with the 3 Category Hedonic Scale. After sufficient numbness is achieved, local infiltrative injection will be performed. Anxiety levels will be evaluated by measuring with the same parameters before topical anaesthesia application, during topical anaesthesia application and injection.
  Interventions: Drug: Topical anesthetic gel
- Cryotherapy as Distilled Water (Experimental): As cryotherapy material, distilled water solution will be cooled in the refrigerator at +4 degrees, removed from the refrigerator just before the application and a cotton swab will be wetted with this solution and applied to the area. The taste/odour evaluation of the applied topical anaesthetic material will be measured with 3 Category Hedonic Scale. After sufficient numbness is achieved, local infiltrative injection will be performed. Anxiety levels will be evaluated by measuring with the same parameters before, during and after topical anaesthesia application and injection.
  Interventions: Drug: Cryotherapy
- Cryotherapy as Anesthetic Solution (Experimental): The topical anaesthetic solution will be stored in the refrigerator at +4 degrees Celsius, removed from the refrigerator just before the application and a cotton swab will be wetted with this solution and applied to the area. The taste/odour evaluation of the applied topical anaesthetic material will be measured with 3 Category Hedonic Scale. After sufficient numbness is achieved, local infiltrative injection will be performed. Anxiety levels will be evaluated by measuring with the same parameters before, during and after topical anaesthesia application and injection.
  Interventions: Drug: Cryotherapy; Drug: topical anesthetic

INTERVENTIONS:
Drug: Cryotherapy — Using crytotherapy as topical anesthetic
  Arms: Cryotherapy as Anesthetic Solution; Cryotherapy as Distilled Water
Drug: topical anesthetic — Comparing the two versions (the room temperature and + 4°C) of the gold standard of local anesthetics, the solution, which contains lidocaine.
  Arms: Cryotherapy as Anesthetic Solution; Topical Anesthetic Solution
Drug: Topical anesthetic gel — Tolerable taste, containing benzocaine at gel formula.
  Arms: Topical Anesthetic Gel

SUMMARY:
In this study, the investigators aimed to compare the effects of topical anesthetic materials and cold application on pain perception. The main questions it aims to answer are:

* Is cold application is effective as a topical anesthetic replacement?
* Is there a difference on pain perception between cold and room temperature topical anesthetic?

The treatment contains of participants selected from a group of patients who requires dental treatment. The mission of the participants is to answer the questionnaires correctly and cooperate the treatment. Participants will be divided into 4 groups containing 25 child per group:

* First group: topical anesthetic spray solution.
* Second group: topical anesthetic gel
* Third group: Cryotherapy as distilled water
* Fourth group: Cryotherapy as topical anesthetic spray solution. All participants will answer questionnaire of pain, anxiety and taste. The oxygen saturation and pulses will be measured with a pulse-oxymeter device to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 10 years old,
* Literate,
* ASA score 1 and 2,
* FRANKL score 3 and 4
* Modified Dental Anxiety score less than 19,
* Not allergic to the active ingredient of the topical anaesthetics used
* Indication for treatment of primary teeth,
* Children who have never had dental treatment under local anaesthesia,
* Patients who agree to participate in the study will be included in the study

Exclusion Criteria:

* Not between the ages of 7 and 10,
* Illiterate,
* ASA score greater than 2,
* FRANKL score 1 and 2
* Modified Dental Anxiety score greater than 19,
* Known allergy to the active ingredient of the topical anaesthetics used
* Children with previous dental experience will not be included in the study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Eased Injection Pain | From the beginning of the topical anesthetic implementation to the injection
  During the procedure, all of the data of the participants containing oxygen saturation, pulse and questionnaire about their experience will be collected to assess the statistical differences between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Faculty of Dentistry, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee HS. Recent advances in topical anesthesia. J Dent Anesth Pain Med. 2016 Dec;16(4):237-244. doi: 10.17245/jdapm.2016.16.4.237. Epub 2016 Dec 31. PMID 28879311
- [Background] Kravitz ND. The use of compound topical anesthetics: a review. J Am Dent Assoc. 2007 Oct;138(10):1333-9; quiz 1382. doi: 10.14219/jada.archive.2007.0048. PMID 17908846
- [Background] Kwiecien SY, McHugh MP. The cold truth: the role of cryotherapy in the treatment of injury and recovery from exercise. Eur J Appl Physiol. 2021 Aug;121(8):2125-2142. doi: 10.1007/s00421-021-04683-8. Epub 2021 Apr 20. PMID 33877402
- [Background] Garcia C, Karri J, Zacharias NA, Abd-Elsayed A. Use of Cryotherapy for Managing Chronic Pain: An Evidence-Based Narrative. Pain Ther. 2021 Jun;10(1):81-100. doi: 10.1007/s40122-020-00225-w. Epub 2020 Dec 14. PMID 33315183
- [Background] Malanga GA, Yan N, Stark J. Mechanisms and efficacy of heat and cold therapies for musculoskeletal injury. Postgrad Med. 2015 Jan;127(1):57-65. doi: 10.1080/00325481.2015.992719. Epub 2014 Dec 15. PMID 25526231
- [Background] Nadler SF, Weingand K, Kruse RJ. The physiologic basis and clinical applications of cryotherapy and thermotherapy for the pain practitioner. Pain Physician. 2004 Jul;7(3):395-9. PMID 16858479
- [Background] Ghaderi F, Banakar S, Rostami S. Effect of pre-cooling injection site on pain perception in pediatric dentistry: "A randomized clinical trial". Dent Res J (Isfahan). 2013 Nov;10(6):790-4. PMID 24379869
- [Background] Lakshmanan L, Ravindran V. Efficacy of Cryotherapy Application on the Pain Perception during Intraoral Injection: A Randomized Controlled Trial. Int J Clin Pediatr Dent. 2021 Sep-Oct;14(5):616-620. doi: 10.5005/jp-journals-10005-2032. PMID 34934271